CLINICAL TRIAL: NCT00379002
Title: The Women's Urology Center/WISH Database Project
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Principal Investigator, Corewell Health East
Other Study IDs: 2006-095
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Interstitial Cystitis; Sexual Dysfunction; Pelvic Pain; Incontinence
Keywords: Interstitial Cystitis; Sexual Dysfunction; Vulvodynia; Pelvic Pain; incontinence
MeSH Terms: conditions — Cystitis, Interstitial; Sexual Dysfunction, Physiological; Pelvic Pain; Vulvodynia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comprehensive database from the Women's Urology Center/WISH (Women's Initiative for Pelvic Pain and Sexual Health) program at Beaumont.

DETAILED DESCRIPTION:
This women's health database will help us to identify health issues/concerns, useful therapies and interventions, and identify areas for improvement or further research specific for women's health. It will allow evaluation of outcomes of clinical interventions to enhance the care and treatment of women with pelvic pain and sexual health concerns.

ELIGIBILITY:
Inclusion Criteria:

All Women's Urology Center or WISH patients will be included in this database over time.

Exclusion Criteria:

The only exclusion would be if specified by a patient upon consent to treatment in the Women's Urology Center or WISH program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Women's Urology Center or WISH patients
Sampling Method: Non-Probability Sample
Enrollment: 2923 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — William Beaumont Hospital Royal Oak
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No